CLINICAL TRIAL: NCT07287137
Title: IDCRP-154: Comparative Immunogenicity of Respiratory Virus Vaccines (CIRV2) Study
Brief Title: Comparative Immunogenicity of Respiratory Virus Vaccines (CIRV2) Study
Acronym: CIRV2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); U.S. Food and Drug Administration (FDA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDCRP-154
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: COVID -19; COVID - 19; COVID 19; Influenza; Respiratory Virus; Respiratory Viruses; Respiratory Virus Infection; Respiratory Virus Infections
Keywords: COVID-19 vaccine; Influenza vaccine; Respiratory virus vaccine; Immunogenicity
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Intervention Model Description: Enrollment of 50-54 individuals to receive the vaccine (up to 27 per arm) per year.
Masking Description: Open-label, with concealment of vaccine allocation until time of vaccination and blinding of all laboratory personnel conducting antibody assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- For fall of 2025, Arm 1 of the study will be the Pfizer-BioNTech mRNA COVID-19 vac (Active Comparator): Arm 1 of the study will be Pfizer-BioNTech mRNA COVID-19 vaccine
  Interventions: Drug: Pfizer-BioNTech mRNA COVID-19 vaccine
- For fall of 2025, Arm 2 of the study will be the Novavax recombinant protein vaccine (Active Comparator): Arm 2 of the study will be the Novavax recombinant protein vaccine
  Interventions: Drug: Novavax recombinant protein vaccine

INTERVENTIONS:
Drug: Pfizer-BioNTech mRNA COVID-19 vaccine — COVID-19 Vaccine, mRNA
  Arms: For fall of 2025, Arm 1 of the study will be the Pfizer-BioNTech mRNA COVID-19 vac
Drug: Novavax recombinant protein vaccine — Recombinant protein vaccine
  Arms: For fall of 2025, Arm 2 of the study will be the Novavax recombinant protein vaccine

SUMMARY:
CIRV2 is a Phase IV randomized, open-label, trial of FDA-approved COVID-19 and/or influenza vaccines (no more than minimal risk) with longitudinal follow-up. In 2025 CIRV2 will compare immunogenicity and reactogenicity of the recombinant Novavax COVID-19 vaccine and the mRNA Pfizer-BioNTech COVID-19 vaccine.

DETAILED DESCRIPTION:
The goal of the Comparative Immunogenicity of Respiratory Virus Vaccines (CIRV2) study is to conduct, on a yearly basis, direct comparisons of immunogenicity and reactogenicity of the most recent versions of FDA-approved vaccines for COVID-19 and/or influenza. Studies will be conducted on individuals that are FDA eligible to receive these vaccines and do not have a medical condition that severely impairs their immune system. For 2025, the study will directly compare the immunogenicity and reactogenicity of the 2025 Novavax recombinant COVID-19 vaccine with the 2025 Pfizer/BioNTech mRNA COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria

1. 18-79 years old
2. Have a history of any of the following risk factors for severe COVID:

   * Asthma
   * Physical inactivity (defined as <150 mins of moderate activity per week or <75 mins of vigorous activity per week)
   * HIV with CD4 count ≥ 500 cells/ul
   * Current or prior smoker
   * Depression or other mood disorder
   * Schizophrenia spectrum disorder
   * Cerebrovascular disease
   * Heart failure
   * Coronary artery disease
   * Cardiomyopathy
   * Pulmonary embolism
   * Pulmonary hypertension
   * Cystic fibrosis
   * Bronchiectasis
   * Chronic obstructive pulmonary disease
   * Interstitial Lung Disease
   * Stage I or II chronic kidney disease
   * Stage 1 defined as normal GFR (> 90) but with other signs of kidney damage such as proteinuria or hematuria
   * Stage 2 defined as having a glomerular filtration rate (GFR) of 60 - 89 ml/min/1.73m2
   * Gestational diabetes
   * Type 1 diabetes with most recent HgbA1C < 7.5%
   * Type 2 diabetes with most recent HgbA1C < 7.5%
   * Obesity with BMI ≥ 30 and < 40
   * Liver disease without cirrhosis and with liver enzyme levels
   * (AST and ALT) no greater than three times the upper limit of normal
3. Military Health System beneficiary and DEERS eligible
4. Willing to be randomized to receive either the Novavax COVID-19 vaccine or the mRNA Pfizer-BioNTech COVID-19 vaccine
5. Will be able to return for a clinic visit in approximately 30 days and be able to follow-up online for the next 9 months.

Exclusion Criteria

1. History of severe allergy or severe adverse reaction such as myocardial inflammation to any component of the mRNA COVID-19 vaccines or the Novavax recombinant COVID-19 vaccine
2. Received a COVID-19 vaccine in the last 3 months.
3. Tested positive for COVID-19 in the past 3 months.

   - Presence of fever, cough, chills, shortness of breath, runny nose, or sore throat today on day of screening/enrollment visit.
4. Active use of immune modulating medications.

   - Defined as active use of chronic immune modulating medications such as systemic corticosteroids at a dose equivalence of 20 mg prednisone or greater daily for over one month, chemotherapy, cytokine inhibitors, or agents that reduce T cell or B cell numbers or function.
5. Diagnosed with immunocompromised stated.

   - Defined as: presence of a disease that is actively causing severe immune suppression or history of prior splenectomy (removal of spleen).
6. Diabetes with the most recent HgbA1C ≥ 7.5.
7. Stage III or greater chronic kidney disease

   - Defined as estimated glomerular filtration rate < 60 ml/min/1.73m2)
8. Obesity with a BMI ≥ 40
9. HIV with a CD4 cell count < 500 cells/ul
10. History of solid organ or bone marrow transplant.
11. Active malignancy

    - Defined as any cancer that is currently being treated or has shown evidence of progression within the past year.
12. Chronic liver disease with compensated or decompensated cirrhosis, or liver enzyme levels (AST or ALT) greater than three times the upper limit of normal.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Variant-specific immune responses | IgG binding antibody levels and neutralizing antibody titers will be assessed on serum samples obtained just prior to vaccination and 30 days (+/- 10 days) after vaccination.
  The primary endpoint is variant-specific immune response (magnitude and breadth) to licensed recombinant and mRNA COVID-19 products administered to healthy adult MHS beneficiaries. This will include quantifying the magnitude of binding and neutralizing antibodies to the vaccine variants and to the dominant variant present one month post-vaccination. Specifically, we will test neutralizing titers (defined as the inverse serum dilution causing a 50% reduction in relative light units in a pseudovirus neutralization assay) and IgG binding antibody levels (measured in arbitrary units) against the following SARS-CoV-2 variants: NB.1.8.1 and XFG (predominant circulating strains in fall 2025), JN.1 and LP.8.1 (vaccine strains), and Wuhan-1 (ancestral strain).

OTHER OUTCOMES:
Vaccine reactogenicity and other incident adverse events (compared between two licensed COVID-19 platforms - recombinant and mRNA) | Reactogenicity and other incident adverse events will be assessed through 9 months after vaccination.
  For vaccine reactogenicity and other incident adverse events, we will use Fisher exact test or a Chi-square test between study arms. Any comparisons among substrata (e.g., age strata, infection histories) will use multiplicity adjustment.
Frequency of participant-reported test positive (antigen and/or PCR) SARS-CoV-2 infections (compared between two licensed COVID-19 platforms - recombinant and mRNA) during the eight months following COVID vaccination and assessment of their symptom patte | Through 9 months after vaccination.
  Frequency of participant-reported test positive infections during the eight months following COVID-19 vaccination will be compared using Fisher exact test or a Chi-square test between study arms. Any comparisons among substrata (e.g., age strata, infection histories) will use multiplicity adjustment.
  Frequency of self-reported COVID-19 symptom severity (% with moderate or greater severity), and duration of illness (in days), will be compared using Fisher exact test or a Chi-square test between study arms. Any comparisons among substrata (e.g., age strata, infection histories) will use multiplicity adjustment.
Salivary and nasopharyngeal IgG and IgA antibody levels to vaccine SARS-CoV-2 strain and dominant SARS-CoV-2 circulating strain at 30 days post vaccination | These antibody tests will be conducted on biosamples obtained just prior to vaccination and 30 days (+/- 10 days) after vaccination.
  Salivary and nasopharyngeal IgG and IgA antibody levels to vaccine SARS-CoV-2 strain and dominant SARS-CoV-2 circulating strain at 30 days post vaccination will be compared between the study arms using GMT and GSD. T-tests will compare responses across two SARS-CoV-2 variants (i.e., the vaccine variant and the dominant circulating variant at the time of vaccination), stratified by vaccine type and adjusted for multiple comparisons (e.g., a Tukey's adjustment). A non-parametric comparison can be used if there is non-normally distributed data despite the use of GMT, these approaches also account for multiplicity (e.g., Kruskall-Wallis with a Dunn's adjustment for multiplicity adjustment).
Antigenic cartography and antibody landscapes | Antigenic cartography studies may be conducted using neutralizing antibody titers obtained just prior to vaccination and 30 days (+/- 10 days) after vaccination.
  Antigenic cartography and antibody landscapes may be performed by FDA collaborators to visualize antigenic drift from the vaccine with sequential variants, leveraging prior analysis approaches used by the study team. These analyses use relative differences in neutralizing antibody responses to generate two-dimensional maps (antigenic cartography) or three-dimensional landscapes that enable one to assess how antigenically similar different virus strains are to each other. Antibody landscapes are useful tools which can capture differential multiple serial antigenic exposures in comparisons of antibody titer and breadth between individuals assigned to receive the recombinant or mRNA vaccines (see examples from Wang et al., Cell Host Microbe, 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Edward Mitre, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] McLeod C, Dymock M, Flanagan KL, Plebanski M, Marshall H, Estcourt MJ, Tjiam MC, Blyth CC, Subbarao K, Mordant FL, Nicholson S, Faust SN, Wadia U, Thornton RB, Ellis Z, Mckenzie A, Marsh JA, Snelling TL, Richmond P. The Platform Trial In COVID-19 Priming and BOOsting (PICOBOO): The immunogenicity, reactogenicity, and safety of different COVID-19 vaccinations administered as a second booster (fourth dose) in AZD1222 primed individuals aged 50-<70 years old. J Infect. 2024 Dec;89(6):106286. doi: 10.1016/j.jinf.2024.106286. Epub 2024 Sep 26. PMID 39341401
- [Background] National Center for Advancing Translational Sciences. Serious adverse events. Available at ht tps://toolkit.ncats.nih.gov/glossary/serious-adverse-event/; accessed 2 January 2025.
- [Background] Wang W, Lusvarghi S, Subramanian R, Epsi NJ, Wang R, Goguet E, Fries AC, Echegaray F, Vassell R, Coggins SA, Richard SA, Lindholm DA, Mende K, Ewers EC, Larson DT, Colombo RE, Colombo CJ, Joseph JO, Rozman JS, Smith A, Lalani T, Berjohn CM, Maves RC, Jones MU, Mody R, Huprikar N, Livezey J, Saunders D, Hollis-Perry M, Wang G, Ganesan A, Simons MP, Broder CC, Tribble DR, Laing ED, Agan BK, Burgess TH, Mitre E, Pollett SD, Katzelnick LC, Weiss CD. Antigenic cartography of well-characterized human sera shows SARS-CoV-2 neutralization differences based on infection and vaccination history. Cell Host Microbe. 2022 Dec 14;30(12):1745-1758.e7. doi: 10.1016/j.chom.2022.10.012. Epub 2022 Oct 21. PMID 36356586
- [Background] Wang W, Bhushan G, Paz S, Stauft CB, Selvaraj P, Goguet E, Bishop-Lilly KA, Subramanian R, Vassell R, Lusvarghi S, Cong Y, Agan B, Richard SA, Epsi NJ, Fries A, Fung CK, Conte MA, Holbrook MR, Wang TT, Burgess TH, Pollett SD, Mitre E, Katzelnick LC, Weiss CD. Human and hamster sera correlate well in identifying antigenic drift among SARS-CoV-2 variants, including JN.1. J Virol. 2024 Nov 19;98(11):e0094824. doi: 10.1128/jvi.00948-24. Epub 2024 Oct 4. PMID 39365051
- [Background] Conner TL, Goguet E, Haines-Hull H, et al: Subclinical SARS-CoV-2 Infections and Endemic Human Coronavirus Immunity Shape SARS-CoV-2 Saliva Antibody Responses. MedRxiv 2024; doi .org/10.1101/2024.05.22.24307751.
- [Background] Laing ED, Weiss CD, Samuels EC, Coggins SA, Wang W, Wang R, Vassell R, Sterling SL, Tso MS, Conner T, Goguet E, Moser M, Jackson-Thompson BM, Illinik L, Davies J, Ortega O, Parmelee E, Hollis-Perry M, Maiolatesi SE, Wang G, Ramsey KF, Reyes AE, Alcorta Y, Wong MA, Lindrose AR, Duplessis CA, Tribble DR, Malloy AMW, Burgess TH, Pollett SD, Olsen CH, Broder CC, Mitre E. Durability of Antibody Response and Frequency of SARS-CoV-2 Infection 6 Months after COVID-19 Vaccination in Healthcare Workers. Emerg Infect Dis. 2022 Apr;28(4):828-832. doi: 10.3201/eid2804.212037. Epub 2022 Feb 24. PMID 35203111
- [Background] Jackson-Thompson BM, Goguet E, Laing ED, Olsen CH, Pollett S, Hollis-Perry KM, Maiolatesi SE, Illinik L, Ramsey KF, Reyes AE, Alcorta Y, Wong MA, Davies J, Ortega O, Parmelee E, Lindrose AR, Moser M, Graydon E, Letizia AG, Duplessis CA, Ganesan A, Pratt KP, Malloy AM, Scott DW, Anderson SK, Snow AL, Dalgard CL, Powers JH 3rd, Tribble D, Burgess TH, Broder CC, Mitre E. Prospective Assessment of SARS-CoV-2 Seroconversion (PASS) study: an observational cohort study of SARS-CoV-2 infection and vaccination in healthcare workers. BMC Infect Dis. 2021 Jun 9;21(1):544. doi: 10.1186/s12879-021-06233-1. PMID 34107889
- [Background] U.S. Food and Drug Administration. Highlights of prescribing information: COMIRNATY® (COVID-19 Vaccine, mRNA) suspension for injection, for intramuscular use. 2024. Available at ht tps://www.fda.gov/media/151707/download; accessed 2 January 2025.
- [Background] U.S. Food and Drug Administration. Fact Sheet for healthcare providers administering vaccine: Emergency Use Authorization of Novavax COVID-19 Vaccine, adjuvanted (2024 - 2025 formula), for individuals 12 years of age and older. 2024. Available at https://www.fda.gov /media/159897/download; accessed 2 January 2025.
- [Background] Fong Y, Huang Y, Benkeser D, Carpp LN, Anez G, Woo W, McGarry A, Dunkle LM, Cho I, Houchens CR, Martins K, Jayashankar L, Castellino F, Petropoulos CJ, Leith A, Haugaard D, Webb B, Lu Y, Yu C, Borate B, van der Laan LWP, Hejazi NS, Randhawa AK, Andrasik MP, Kublin JG, Hutter J, Keshtkar-Jahromi M, Beresnev TH, Corey L, Neuzil KM, Follmann D, Ake JA, Gay CL, Kotloff KL, Koup RA, Donis RO, Gilbert PB; Immune Assays Team; Coronavirus Vaccine Prevention Network (CoVPN)/2019nCoV-301 Principal Investigators and Study Team; United States Government (USG)/CoVPN Biostatistics Team. Immune correlates analysis of the PREVENT-19 COVID-19 vaccine efficacy clinical trial. Nat Commun. 2023 Jan 19;14(1):331. doi: 10.1038/s41467-022-35768-3. PMID 36658109
- [Background] Weitzman ER, Sherman AC, Levy O. SARS-CoV-2 mRNA Vaccine Attitudes as Expressed in U.S. FDA Public Commentary: Need for a Public-Private Partnership in a Learning Immunization System. Front Public Health. 2021 Jul 16;9:695807. doi: 10.3389/fpubh.2021.695807. eCollection 2021. PMID 34336774
- [Background] Biggs AT, Littlejohn LF. Describing mRNA Vaccine Technology for a Military Audience. Mil Med. 2023 Mar 20;188(3-4):547-554. doi: 10.1093/milmed/usac129. PMID 35584186
- [Background] Marchese AM, Rousculp M, Macbeth J, Beyhaghi H, Seet BT, Toback S. The Novavax Heterologous Coronavirus Disease 2019 Booster Demonstrates Lower Reactogenicity Than Messenger RNA: A Targeted Review. J Infect Dis. 2024 Aug 16;230(2):e496-e502. doi: 10.1093/infdis/jiad519. PMID 37992183
- [Background] Scher AI, Berjohn CM, Byrne C, Colombo RE, Colombo CJ, Edwards MS, Ewers EC, Ganesan A, Jones M, Larson DT, Libraty D, Lindholm DA, Madar CS, Maldonado CJ, Maves RC, Mende K, Richard SA, Rozman JS, Rusiecki J, Smith A, Simons M, Tribble D, Agan B, Burgess TH, Pollett SD; EPICC COVID-19 Cohort Study Group. An Analysis of SARS-CoV-2 Vaccine Reactogenicity: Variation by Type, Dose, and History, Severity, and Recency of Prior SARS-CoV-2 Infection. Open Forum Infect Dis. 2022 Jun 28;9(7):ofac314. doi: 10.1093/ofid/ofac314. eCollection 2022 Jul. PMID 35899278
- [Background] U.S. Food and Drug Administration. FDA Briefing Document. Vaccines and Related Biological Products Advisory Committee Meeting June 5, 2024. 2024. Available at https://www.fda.gov /media/179003/download; accessed 10 October 2024.
- [Background] U.S. Food and Drug Administration. Vaccines and Related Biological Products Advisory Committee June 5, 2024 Meeting Announcement. 2024. Available at https://www.fda.gov /advisory-committees/advisory-committee-calendar/vaccines-and-related-biological- products-advisory-committee-june-5-2024-meeting-announcement; accessed 10 October 2024.
- [Background] Winkler EL, Stahlman SL, Wells NY, Chauhan AV, Hiban KM, Costello AA, Mancuso JD. COVID-19 Booster Vaccination in the U.S. Military, August 2021-January 2022. Am J Prev Med. 2023 Feb;64(2):270-274. doi: 10.1016/j.amepre.2022.07.017. Epub 2022 Aug 29. PMID 36123230
- [Background] Centers for Disease Control and Prevention. ACIP Evidence to Recommendations (EtR) for Use of 2024-2025 COVID-19 Vaccines in Persons ≥6 Months of Age. 2024. Available at https:// www.cdc.gov/vaccines/acip/recs/grade/covid-19-2024-2025-6-months-and-older-etr. html; accessed 10 October 2024.
- [Background] Centers for Disease Control and Prevention. Staying Up to Date with COVID-19 Vaccines. 2024. Available at https://www.cdc.gov/covid/vaccines/stay-up-to-date.html; accessed 10 October 2024.
- [Background] Lam ICH, Zhang R, Man KKC, Wong CKH, Chui CSL, Lai FTT, Li X, Chan EWY, Lau CS, Wong ICK, Wan EYF. Persistence in risk and effect of COVID-19 vaccination on long-term health consequences after SARS-CoV-2 infection. Nat Commun. 2024 Feb 26;15(1):1716. doi: 10.1038/s41467-024-45953-1. PMID 38403654
- [Background] Richard SA, Scher AI, Rusiecki J, Byrne C, Berjohn CM, Fries AC, Lalani T, Smith AG, Mody RM, Ganesan A, Huprikar N, Colombo RE, Colombo CJ, Schofield C, Lindholm DA, Mende K, Morris MJ, Jones MU, Flanagan R, Larson DT, Ewers EC, Bazan SE, Saunders D, Maves RC, Livezey J, Maldonado CJ, Edwards MS, Rozman JS, O'Connell RJ, Simons MP, Tribble DR, Agan BK, Burgess TH, Pollett SD; EPICC COVID-19 Cohort Study Group. Decreased Self-reported Physical Fitness Following SARS-CoV-2 Infection and the Impact of Vaccine Boosters in a Cohort Study. Open Forum Infect Dis. 2023 Nov 17;10(12):ofad579. doi: 10.1093/ofid/ofad579. eCollection 2023 Dec. PMID 38130596
- [Background] Hone E, Pollett SD, Richard SA, et al, editors. The Molecular Epidemiology and Congregate Transmission Dynamics of Acute Respiratory Infections (ARIs) at United States Naval Academy (USNA) during Plebe Summer. Poster #113. Military Health System Research Symposium; 2024; Kissimmee, FL.
- [Background] Armed Forces Health Surveillance Division. Absolute and relative morbidity burdens attributable to various illnesses and injuries among active component members of the U.S. Armed Forces, 2023. MSMR. 2024 Jun 20;31(6):2-10. PMID 38981057
- [Background] Armed Forces Health Surveillance Division. Absolute and relative morbidity burdens attributable to various illnesses and injuries among non-service member beneficiaries of the Military Health System, 2023. MSMR. 2024 Jul 20;31(7):11-20. PMID 39136697
- [Background] Taylor CA, Patel K, Pham H, Kirley PD, Kawasaki B, Meek J, Witt L, Ryan PA, Reeg L, Como-Sabetti K, Domen A, Anderson B, Bushey S, Sutton M, Talbot HK, Mendez E, Havers FP; COVID-NET Surveillance Team. COVID-19-Associated Hospitalizations Among U.S. Adults Aged >/=18 Years - COVID-NET, 12 States, October 2023-April 2024. MMWR Morb Mortal Wkly Rep. 2024 Oct 3;73(39):869-875. doi: 10.15585/mmwr.mm7339a2. PMID 39361542
- [Background] National Center for Health Statistics. Provisional COVID-19 Mortality Surveillance. Centers for Disease Control and Prevention; 2024. Available at https://www.cdc.gov/nchs/nvss/vsrr /covid19/index.htm; accessed 10 October 2024.
- [Background] Kasper MR, Geibe JR, Sears CL, Riegodedios AJ, Luse T, Von Thun AM, McGinnis MB, Olson N, Houskamp D, Fenequito R, Burgess TH, Armstrong AW, DeLong G, Hawkins RJ, Gillingham BL. An Outbreak of Covid-19 on an Aircraft Carrier. N Engl J Med. 2020 Dec 17;383(25):2417-2426. doi: 10.1056/NEJMoa2019375. Epub 2020 Nov 11. PMID 33176077
- [Background] Mease LE, Smith AM. Surveillance snapshot: A simple model estimating the impact ofCOVID-19 on lost duty days among U.S. service members. MSMR. 2021 Sep 1;28(9):17. No abstract available. PMID 34854661
- [Background] U.S. Department of Defense. Coronavirus: DoD Response. 2024. Available at https://www. defense.gov/Spotlights/Coronavirus-DOD-Response/; accessed 8 October 2024.
- [Background] Absolute and relative morbidity burdens attributable to various illnesses and injuries, active component, U.S. Armed Forces, 2020. MSMR. 2021 May;28(5):2-9. No abstract available. PMID 34155889
- [Background] Sanchez JL, Cooper MJ, Myers CA, Cummings JF, Vest KG, Russell KL, Sanchez JL, Hiser MJ, Gaydos CA. Respiratory Infections in the U.S. Military: Recent Experience and Control. Clin Microbiol Rev. 2015 Jul;28(3):743-800. doi: 10.1128/CMR.00039-14. PMID 26085551
- [Background] Gray GC, Callahan JD, Hawksworth AW, Fisher CA, Gaydos JC. Respiratory diseases among U.S. military personnel: countering emerging threats. Emerg Infect Dis. 1999 May-Jun;5(3):379-85. doi: 10.3201/eid0503.990308. PMID 10341174